CLINICAL TRIAL: NCT07067424
Title: The Effect of Lavender and Bergamot Aromatherapy Before Colonoscopy on Anxiety, Vital Signs, and Feelings of Embarrassment"
Brief Title: Effect of Aromatherapy on Anxiety in Colonoscopy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, ERAY YÜCEDAĞ, Clinical Nurse, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EY-Aroma2025-01
Record Dates: First submitted 2025-07-14; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Colonoscopy; Aromatherapy
Keywords: Lavender; Bergamot; Anxiety; Colonoscopy; Embarrassment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lavender Aromatherapy (Experimental): Inhalation of lavender essential oil for 20 minutes prior to colonoscopy.
  Interventions: Other: Lavender Aromatherapy
- Bergamot Aromatherapy (Experimental): Inhalation of bergamot essential oil for 20 minutes prior to colonoscopy.
  Interventions: Other: Bergamot Aromatherapy
- Control Group (Placebo Comparator): Participants in this group will inhale an odorless substance (distilled water ) to mimic the aromatherapy procedure without active ingredients.
  Interventions: Other: Placebo Inhalation

INTERVENTIONS:
Other: Lavender Aromatherapy — Participants will inhale lavender essential oil via cotton pads placed near the nose for 20 minutes prior to colonoscopy. The application will take place in a pre-procedure waiting area under nurse supervision.
  Arms: Lavender Aromatherapy
Other: Bergamot Aromatherapy — Participants will inhale bergamot essential oil through cotton pads placed near the nose for 20 minutes before the colonoscopy procedure, under the supervision of clinical staff.
  Arms: Bergamot Aromatherapy
Other: Placebo Inhalation — Participants will inhale an odorless substance (distilled water) using the same method and duration as the intervention groups, to simulate the aromatherapy procedure.
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the effects of aromatherapy with lavender and bergamot essential oils on anxiety, vital signs, and feelings of embarrassment before colonoscopy. The findings of this study are expected to contribute both to filling a gap in the literature and to the planning of evidence-based nursing interventions aimed at minimizing pre-colonoscopy anxiety and embarrassment in patients.

DETAILED DESCRIPTION:
In addition to being a painful and uncomfortable procedure, colonoscopy can cause anxiety and fear in patients due to procedure-related concerns, fear of a cancer diagnosis, and feelings of embarrassment resulting from perceived violations of privacy during the procedure. To alleviate patients' anxiety, fear, or embarrassment before colonoscopy, various non-pharmacological approaches, such as aromatherapy, are utilized. Aromatherapy, also known as essential oil therapy, is defined as "the art and science of using naturally extracted aromatic essences from plants to balance, harmonize, and promote the health of the body, mind, and spirit". Lavender and bergamot essential oils have been reported to have positive effects on anxiety in patients undergoing certain medical procedures, such as surgeries, childbirth, urodynamic testing, and endoscopic interventions. However, no study has yet evaluated the combined effects of aromatherapy with lavender and bergamot oils on anxiety, vital signs, and feelings of embarrassment in patients undergoing colonoscopy. The aim of this study is to investigate the effects of aromatherapy with lavender and bergamot essential oils on anxiety, vital signs, and feelings of embarrassment before colonoscopy. The findings of this study are expected to contribute both to filling a gap in the literature and to the planning of evidence-based nursing interventions aimed at minimizing pre-colonoscopy anxiety and embarrassment in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing a colonoscopy
* Patients capable of reading and understanding the study instructions

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients who reported an allergy to any of the lavender or bergamot extracts used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety level measured by the State Anxiety Inventory (STAI-State) | Immediately before and 30 minutes after the intervention
  Anxiety will be assessed using the State Anxiety Inventory (STAI-State), which consists of 20 items rated on a 4-point Likert scale. The total score ranges from 20 to 80, with higher scores indicating greater anxiety. The scale has been validated in Turkish with a Cronbach's alpha between 0.94 and 0.96.

SECONDARY OUTCOMES:
Change in embarrassment level measured by the Colonoscopy Embarrassment Scale | Immediately after the colonoscopy procedure
  Embarrassment related to colonoscopy will be measured using the 15-item Colonoscopy Embarrassment Scale, with scores ranging from 15 to 60. Higher scores indicate greater embarrassment. The Turkish version has a Cronbach's alpha of 0.94.

OTHER OUTCOMES:
Change in heart rate | Immediately before and 30 minutes after the intervention
  Heart rate (beats per minute) will be measured using a standard monitoring form.
Change in respiratory rate | Immediately before and 30 minutes after the intervention
  Respiratory rate (breaths per minute) will be measured using a standard monitoring form.
Change in systolic and diastolic blood pressure | Immediately before and 30 minutes after the intervention
  Systolic and diastolic blood pressure will be measured in mmHg using a standard blood pressure monitor.
Change in oxygen saturation | Immediately before and 30 minutes after the intervention
  Oxygen saturation (SpO₂) will be measured using pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Eray Yucedag, MSc Student, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Famagusta State Hospital, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yue QQ, Feng GH, Peng T, Tang T, Sun YX, Meng XR, Huang LL, Zhao KH, Huang HL, Zeng Y. What is the current state of anxiety and its related factors in Chinese patients undergoing colonoscopy? A cross-sectional study. BMC Psychol. 2025 Feb 27;13(1):169. doi: 10.1186/s40359-025-02463-z. PMID 40016795
- [Result] Peng W, McKinnon-Crowley J, Huang Q, Mao B. Assessing Fear, Embarrassment, and Disgust in Colonoscopy: The Development of Measurement Instruments and Psychometric Evidence. Health Educ Behav. 2024 Aug;51(4):601-612. doi: 10.1177/10901981231177075. Epub 2023 Jun 9. PMID 37293778
- [Result] Mutlu S, Yilmaz E, Sahin ST. The effect of position change and abdominal massage on anxiety, pain and distension after colonoscopy: A randomized clinical trial. Explore (NY). 2024 Jan-Feb;20(1):89-94. doi: 10.1016/j.explore.2023.06.007. Epub 2023 Jun 20. PMID 37391282
- [Result] Dogan Yilmaz E, Unlusoy Dincer N. The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):318-328. doi: 10.1097/SGA.0000000000000733. Epub 2023 Jun 5. PMID 37278621
- [Result] Honig AJ, Galassi MG, Ogungbe OO, Uranga T, Cuevas DK. Implementation of Aromatherapy, a Nonpharmacological Intervention, to Reduce Anxiety During the Preoperative Period. J Perianesth Nurs. 2023 Apr;38(2):206-212. doi: 10.1016/j.jopan.2022.06.011. Epub 2023 Feb 1. PMID 36732122
- [Result] Kettas Dolek E, Altun Ugras G. The effect of aromatherapy during urodynamic testing on patients anxiety and cortisol levels: A randomized controlled trial. Neurourol Urodyn. 2024 Sep;43(7):1591-1599. doi: 10.1002/nau.25491. Epub 2024 May 15. PMID 38747020
- [Result] Ni CH, Hou WH, Kao CC, Chang ML, Yu LF, Wu CC, Chen C. The anxiolytic effect of aromatherapy on patients awaiting ambulatory surgery: a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:927419. doi: 10.1155/2013/927419. Epub 2013 Dec 17. PMID 24454517
- [Result] Keser E, Baglama SS, Sezer C. The Effect of Reiki and Aromatherapy on Vital Signs, Oxygen Saturation, and Anxiety Level in Patients Undergoing Upper Gastrointestinal Endoscopy: A Randomized Controlled Study. Holist Nurs Pract. 2023 Nov-Dec 01;37(6):337-346. doi: 10.1097/HNP.0000000000000611. PMID 37851350
- [Result] Pasyar N, Rambod M, Araghi F. The effect of bergamot orange essence on anxiety, salivary cortisol, and alpha amylase in patients prior to laparoscopic cholecystectomy: A controlled trial study. Complement Ther Clin Pract. 2020 May;39:101153. doi: 10.1016/j.ctcp.2020.101153. Epub 2020 Mar 21. PMID 32379683
- [Result] Hedigan F, Sheridan H, Sasse A. Benefit of inhalation aromatherapy as a complementary treatment for stress and anxiety in a clinical setting - A systematic review. Complement Ther Clin Pract. 2023 Aug;52:101750. doi: 10.1016/j.ctcp.2023.101750. Epub 2023 Apr 5. PMID 37031643
- [Result] Sayilan S, Sayilan AA, Mert S, Oztekin SD, Baydemir C. The Effect of Precolonoscopy Lavender Inhalation on Patient Anxiety and Comfort: A Randomized, Controlled, Double-Blinded, Single-Center Study. Gastroenterol Nurs. 2023 Sep-Oct 01;46(5):376-385. doi: 10.1097/SGA.0000000000000754. Epub 2023 Jun 8. PMID 37289849
- [Result] Vora LK, Gholap AD, Hatvate NT, Naren P, Khan S, Chavda VP, Balar PC, Gandhi J, Khatri DK. Essential oils for clinical aromatherapy: A comprehensive review. J Ethnopharmacol. 2024 Aug 10;330:118180. doi: 10.1016/j.jep.2024.118180. Epub 2024 Apr 16. PMID 38614262
- [Result] Shirzad M, Nasiri E, Hesamirostami M, Akbari H. The Effect of Lavender on Anxiety and Hemodynamic Status Before Septorhinoplasy and Rhinoplasty. J Perianesth Nurs. 2023 Feb;38(1):45-50. doi: 10.1016/j.jopan.2022.05.067. Epub 2022 Aug 18. PMID 35987997